CLINICAL TRIAL: NCT03722485
Title: Hydromechanical Cleansing With V.A.C. VERAFLO CLEANSE CHOICE™ Dressing and NPWTi-d vs. Collagenase Ointment in the Management of Full-thickness Wounds
Brief Title: Negative Pressure Wound Therapy With Instillation of Saline Solution Versus Collagenase Ointment in Full-thickness Wounds
Acronym: ACCELERATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment challenges and business reasons.
Sponsor: KCI USA, Inc (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCI.CLEANSE.CHOICE.2017.02
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Wounds and Injuries; Wound Healing; Granulation Tissue
MeSH Terms: conditions — Wounds and Injuries | interventions — Collagenases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Negative Pressure Therapy w/ instillation and dwell (NPWTi-d) (Experimental): V.A.C. VeraFlo Cleanse Choice Dressing, V.A.C.Ulta Therapy Unit and saline solution
  Interventions: Device: Negative Pressure Therapy w/ instillation and dwell (NPWTi-d)
- Collagenase Ointment (Active Comparator): Collagenase Ointment
  Interventions: Biological: Collagenase Ointment

INTERVENTIONS:
Device: Negative Pressure Therapy w/ instillation and dwell (NPWTi-d) — Negative Pressure Therapy at -125mmHg for 3.5 hours followed by 10 minute dwell of saline solution for 6-9 days.
  Other Names: V.A.C. VeraFlo Cleanse Choice; V.A.C.Ulta Therapy Unit
  Arms: Negative Pressure Therapy w/ instillation and dwell (NPWTi-d)
Biological: Collagenase Ointment — Collagenase ointment applied daily to the wound and covered with secondary dressing for 6-9 days.
  Arms: Collagenase Ointment

SUMMARY:
Evaluation of wound bed surface area containing clean, healthy viable tissue in full-thickness wounds.

DETAILED DESCRIPTION:
This study evaluates changes in wound bed surface area of clean, healthy viable tissue in subjects with full-thickness wounds using negative pressure wound therapy with instillation of saline solution versus a collagenase ointment.

ELIGIBILITY:
Inclusion Criteria:

The Subject:

1. is anticipated to be hospitalized for the duration of treatment (minimum of 6 days).
2. is ≥ 18 years of age.
3. or their legally authorized representative is able to provide informed consent.
4. has been diagnosed with a wound (eg, chronic, acute, traumatic, or dehisced wounds) and/or ulcer (ie, full- thickness wounds) that meets the following criteria:

   1. total surface area measuring ≥ 16 cm2, including a minimum width of 2 cm (before removal of eschar at the bedside and excluding undermining).
   2. < 20 cm across (edge-to-edge) at any point perpendicular to the wound edges.
5. has, in the opinion of the investigator, no more than 2/3 of the wound bed surface area considered to be clean, healthy, and viable. If eschar is present at baseline, it must be removed by bedside debridement prior to assessing the percentage of clean, healthy, and viable wound bed.
6. has a negative urine or serum pregnancy test at screening (if female and has potential for pregnancy) and is willing to take precautionary measures to prevent pregnancy during the duration of the study (up to 9 days).

Exclusion Criteria:

The Subject:

1. has been diagnosed with malignancy in the wound.
2. has untreated osteomyelitis.
3. has an untreated systemic infection.
4. has active cellulitis in the periwound area.
5. has a known allergy or hypersensitivity to study materials: collagenase ointment, dressing(s), and/or dressing components such as acrylic adhesives or polyurethane.
6. has, in the opinion of the investigator, a clinically significant condition that would impair the Subject's ability to comply with the study procedures.
7. has had radiation directly to the wound area.
8. has been diagnosed with a major vascular deficit limiting arterial inflow to the wound region, as determined by the Investigator's interpretation of the Subject's medical history.
9. has eschar in the wound that cannot be removed by bedside sharp and/or mechanical debridement.
10. is participating in another interventional clinical trial for the duration of the study.
11. has unexplored fistulas in the wound or fistulas in the wound that connect to other body cavities.
12. has a wound with any tunneling present.
13. has inadequate hemostasis at the wound site, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Rush University Medical Center, Chicago, Illinois
  - South Shore Hospital Center for Wound Healing, Weymouth, Massachusetts
  - University of Missouri, Columbia, Missouri
  - Northwell Health System - North Shore University Hospital, Manhasset, New York
  - New York University - Winthrop Hospital, Mineola, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) | Collagenase Ointment
Started | 19 | 25
Completed | 15 | 18
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 2
Not completed — subject discharged prior to study completion | 1 | 5
Not completed — eligibility criteria not met | 2 | 0

BASELINE CHARACTERISTICS:
Population: This is the modified intent-to-treat (ITT) population, which is a subset of all subjects randomized who had no more than 2/3 of the wound bed considered to be clean, healthy, and viable, as well as had an end-point assessment on day 6-9.
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) | Collagenase Ointment | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (14.02) | 67.4 (12.97) | 65.5 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 13 | 16 | 29
Wound Type [Count of Participants; unit: Participants]
  Pressure Ulcer | 11 | 15 | 26
  Venous leg ulcer | 2 | 0 | 2
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in the Percentage of Wound Bed Surface Area (%) Considered Clean, Healthy and Viable From Baseline to Day 6-9 Upon Dressing Removal.
Description: The Absolute Change in the Percentage of Wound bed surface area (cm2) considered to be clean, healthy, and viable from baseline to Day 6-9 upon the final dressing removal.
Time Frame: baseline and 6-9 days of treatment
Population: Modified ITT population
Measure: Mean (Standard Deviation); unit: percent wound clean healthy viable.
Arm/Group | Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) | Collagenase Ointment
Number analyzed (Participants) | 13 | 16
percent wound clean healthy viable. | 27.9 (34.35) | 11.6 (40.52)
Statistical Analysis 1: Comparison: Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) vs Collagenase Ointment; Test type: Superiority; p = 0.2920, Regression, Linear — Confounding variables of image capture techniques, image quality and image analysis noted throughout study conduct prohibits any definitive conclusions to be drawn from this analysis; Test of treatment effect using a generalized linear model with treatment arm, baseline values, and clinical site as factors

2. Secondary Outcome: Percent Change in Total Wound Volume (%) From Baseline to Day 6-9 Upon the Final Dressing Removal.
Description: The percent change in total wound volume (%) from baseline to Day 6-9 upon the final dressing removal.
Time Frame: baseline and 6-9 days of treatment
Population: Modified ITT population
Measure: Mean (Standard Deviation); unit: percent change in wound volume
Arm/Group | Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) | Collagenase Ointment
Number analyzed (Participants) | 13 | 16
percent change in wound volume | -0.3 (0.59) | 1.3 (3.27)
Statistical Analysis 1: Comparison: Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) vs Collagenase Ointment; Test type: Superiority; p = 0.0213, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percent Change in Total Wound Area (%) From Baseline to Day 6-9 Upon the Final Dressing Removal.
Description: The percent change in total wound area (%) from baseline to Day 6-9 upon the final dressing removal.
Time Frame: baseline and 6-9 days of treatment
Population: Modified ITT population
Measure: Mean (Standard Deviation); unit: percent change in wound area
Arm/Group | Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) | Collagenase Ointment
Number analyzed (Participants) | 13 | 16
percent change in wound area | 0 (0.20) | 0.1 (0.96)
Statistical Analysis 1: Comparison: Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) vs Collagenase Ointment; Test type: Superiority; p = 0.7422, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Physician Assessment of Need for Wound Debridement
Description: Physician assessment of the need for surgical debridement upon completion of study treatment up to Day 6-9.
Time Frame: 6-9 days of treatment
Population: Modified ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) | Collagenase Ointment
Number analyzed (Participants) | 13 | 16
Participants
  Not needing debridement | 3 | 2
  Yes, needing debridement | 10 | 14
Statistical Analysis 1: Comparison: Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) vs Collagenase Ointment; Test type: Superiority; p = 0.6322, Fisher Exact

ADVERSE EVENTS:
Time Frame: Up to the last study visit, which was labeled as being the 6 to 9-day visit
Description: The safety set consisted of 17 subjects in the Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) group/arm and not 19 subjects (the total randomized to this group/arm) because two subjects were deemed to not meet eligibility criteria post-randomization and did to not receive treatment.
Arm/Group | Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) | Collagenase Ointment
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/17 | 2/25
Other Adverse Events (participants affected / at risk) | 8/17 | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) (N=17) | Collagenase Ointment (N=25)
impaired healing (General disorders) | 1 | 0
sepsis (Infections and infestations) | 1 | 0
post-procedural hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Negative Pressure Therapy w/ Instillation and Dwell (NPWTi-d) (N=17) | Collagenase Ointment (N=25)
fluid overload (Cardiac disorders) | 1 | 0
gastro-intestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 2 | 0
pyrexia (General disorders) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
blood potassium increase (Investigations) | 1 | 0
hemoglobin decrease (Investigations) | 4 | 1
hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
hypotension (Vascular disorders) | 0 | 2
splenic infarction (Blood and lymphatic system disorders) | 0 | 1
atrial fibrillation (Cardiac disorders) | 0 | 1
conjunctivitis (Eye disorders) | 0 | 1
dysphagia (Gastrointestinal disorders) | 0 | 1
epi-gastric discomfort (Gastrointestinal disorders) | 0 | 1
flatulence (Gastrointestinal disorders) | 0 | 1
lethargy (General disorders) | 0 | 1
mucosal hypertrophy (General disorders) | 0 | 1
pain (General disorders) | 0 | 1
candida infection (Infections and infestations) | 0 | 1
osteomyelitis (Infections and infestations) | 0 | 1
wound infection (Infections and infestations) | 0 | 2
blood glucose decreased (Investigations) | 0 | 1
white blood cell count increased (Investigations) | 0 | 1
hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
hyper natremia (Metabolism and nutrition disorders) | 0 | 1
hypokalemia (Metabolism and nutrition disorders) | 0 | 1
hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
device occlusion (Product Issues) | 0 | 1
anxiety (Psychiatric disorders) | 0 | 1
incontinence (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT03722485/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT03722485/SAP_001.pdf